## **Cover Page**

 $Study\ Title: PRescribing\ Interventions\ for\ Chronic\ pain\ using\ the\ Electronic\ Health\ record\ (PRINCE)$ 

ClinicalTrials.gov #: NCT04601506

Consent Form for PDMP Data Access

Document date: November 18, 2020

Dear [primary care clinician],

Fairview and University of Minnesota Physicians are working with researchers at the University of Minnesota to assess the best ways to support opioid prescribing and pain treatment in primary care.

As part of this research, we are asking for you to grant permission to the Minnesota Prescription Monitoring Program (MN PMP) to release to the research team at the University of Minnesota information regarding how often you, or your authorized delegates, have searched the MN PMP database between August 2019-September 2021. By granting your permission, you will help to improve the design of EHR-based tools to support safe and effective opioid prescribing, which can improve the process of care delivery for clinicians and quality of care for patients.

## What we are requesting:

-Your permission to release data on the number of times you and your delegates search the Minnesota PMP.

## What we are not requesting:

- -Any patient-level information.
- -Any information about the reason or clinical content of a PMP query. We only are counting the frequency of searching the PMP.
- -Permission to report any information about specific clinicians or clinics. Any results that are reported will <u>not</u> be able to identify clinicians or even specific clinics.

We do not foresee any potential risks or discomfort to you by allowing the research team to access this information. The records of this study will be kept private. In any sort of report we might publish, we will not include any information that will make it possible to identify any person or clinic. Research records will be stored securely and only researchers will have access to the records. Once all of the data are collected, all personal identifiers will be removed.

Your permission to grant access to this information helps Fairview, University of Minnesota Physicians, and the state of Minnesota to make decisions about how to invest most effectively in resources to support safe and effective pain treatment.

If you have any questions about this research, you can contact Ezra Golberstein at the Division of Health Policy and Management of the University of Minnesota School of Public Health, at 612-626-2572, or email <a href="mailto:egolber@umn.edu">egolber@umn.edu</a>. You may also contact Dr. Brent Elert (<a href="mailto:belert1@fairview.org">belert1@fairview.org</a>), or the Project Manager Ms. Alex Hanson at 612-672-2308 or <a href="mailto:ahanso25@fairview.org">ahanso25@fairview.org</a>.

This research has been reviewed and approved by an IRB within the University of Minnesota Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research

experience, call the Research Participants' Advocate Line at 612-625-1650 (Toll Free: 1-888-224-8636) or go to <u>z.umn.edu/participants</u>.

By signing electronically below, you grant permission to the MN PMP to release to the University of Minnesota Research team the number of times you, or your authorized delegates, have searched the Minnesota PMP database between August 2019-September 2021.

Revocation of this authorization may be done at any time by submitting a request in writing to <a href="minnesota.pmp@state.mn.us">minnesota.pmp@state.mn.us</a>. Thank you for your help on this important project,

| Brent Elert/David Satin | |
|-------------------------|-------------|
| Ezra Golberstein | |
| | <del></del> |
| Signature | Date |